CLINICAL TRIAL: NCT01279889
Title: Predicting Hypotension Resistant to Phenylephrine (PE) Infusion in Elective Cesarean Delivery (CD)
Brief Title: Predicting Hypotension Related to Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Other Study IDs: H10-03231
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Hypotension
Keywords: hypotension; cesarean delivery; cardiac output; blood pressure; plethysmography variability index
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cesarean Delivery: Healthy pregnant women having an elective cesarean delivery

SUMMARY:
This study aims to identify women at risk of low blood pressure (hypotension) after the usual cesarean anesthetic - a spinal anesthetic. Hypotension may be caused by dehydration. We believe we can predict who will get hypotension by using two anesthesia monitors together with a passive leg raise (PLR) (legs elevated after a period spent reclining). The PLR will cause a shift of blood from the legs to the heart, and the monitors will detect the heart's response to tell if a subject is dehydrated. We want to see if these dehydration tests can also predict hypotension after a spinal anesthetic.

DETAILED DESCRIPTION:
We aim to predict the development of spinal anesthesia related hypotension in subjects already receiving a prophylactic infusion of phenylephrine (PE) who are having a cesarean delivery (CD). Hypotension arising in this fashion may signify that a subject is actually relatively fluid-deplete, and might benefit from intravenous (IV) fluid replacement. We will observe the association between hypotension and results of pre-anesthesia tests with two non-invasive monitors used in conjunction with a dynamic cardiovascular fluid challenge (by using a passive leg raise (PLR) maneuver). The use of any therapeutic intervention such as a fluid infusion would be the object of a subsequent study.

We propose that a minority of parturients present for elective CD being relatively fluid deplete. It is our hypothesis that the characteristics of passive leg raise (PLR) induced changes in the plethysmography variability index (PVI generated by the Masimo Radical 7™) and cardiac output (CO as derived from the Non Invasive Cardiac Output Monitor (NICOM) produced by Cheetah Medical™) will identify these subjects and that without large volume fluid administration they are likely to develop hypotension despite the use of a prophylactic PE infusion

Justification: Hypotension is the most common cause of spinal anesthesia related morbidity in cesarean delivery. Hypotension is very common and without treatment can affect over 80% of women. The mechanism is usually twofold: Firstly preload to the right ventricle (RV) is reduced as a result of venodilation from spinal sympathetic blockade. Unfortunately attempting to improve preload by infusion of IV fluid alone doesn't make much difference to the rates of hypotension (only 16% reduction in one large study). The second mechanism results from afterload reduction through arterial vasodilation which directly causes a reduction in blood pressure (BP). The treatment for this is most commonly a PE infusion, and when used this makes a significant difference reducing rates by over 50%. Unfortunately again there are a few who don't seem to respond (the residual of hypotension remains about 30%). Increasing the doses of PE only increases the rate of side effects, without affecting hypotension rates. However, giving both fluid and a PE infusion does seem to prevent hypotension in almost all subjects, suggesting that those who were resistant to PE alone actually did need some fluid. These subjects however are the exception not the rule, and giving fluid to these relatively "fluid deplete" as well as the rest may result in an increase in fluid related side effects. We believe that fluid therapy could be tailored better if we could identify which subjects are actually fluid deplete in the first instance.

Testing to predict fluid responsiveness has been studied in the intensive care unit (ICU) but not in obstetric subjects. Using a PLR increases the return of blood to the right ventricle (RV). In a fluid deplete individual this significantly improves venous return such that CO changes dramatically. In a well hydrated individual venous return is already adequate so the change in CO is less. The NICOM will directly detect the CO change induced by a PLR. The Masimo detects variations in the pulse oximetry plethysmograph trace that result from subtle variations in the cardiac output caused by changes in the intrathoracic pressure from breathing. Intrathoracic pressure increases during expiration in a spontaneously breathing subject and causes a reduction in venous return to the RV which causes a subsequent fall in CO. The variation in the plethysmography signal with respiration is displayed as a percentage index of the baseline signal strength which correlates with how much venous return to the RV is affected by respiration. If a subject's preload is low the plethysmography variability index (PVI) will be high from the dramatic fluctuation in CO with changes in intrathoracic pressure. Unfortunately with spontaneously breathing subjects this value is not consistent enough between individuals for PVI itself to give an accurate indication of fluid volume state. However changes induced in the PVI within an individual subject from a challenge such as fluid infusion or a PLR appear to be better at indicating fluid responsiveness.

We plan to use both the NICOM and the Masimo in conjunction with a PLR to assess fluid state (deplete or otherwise) preoperatively. We will then observe whether or not the pre-anesthesia testing correlates with development of PE infusion resistant hypotension during the routine spinal anesthetic.

The primary objective of this study is to correlate the results of pre-anesthesia testing with actual development of PE infusion resistant hypotension. Secondary outcomes are discussed in statistical analysis below.

ELIGIBILITY:
Inclusion Criteria:

* Height less than 150cm or greater than 180cm
* Body Mass Index (BMI) greater than 40kg/m2: obesity makes accurate non-invasive blood pressure (BP) measurement difficult. It may also affect speed of onset and height of subarachnoid block due to increased epidural venous plexus engorgement and thecal sac compression resulting in more marked hypotension.
* Pregnancy induced hypertension (BP after 20wk greater than 140/90 with proteinuria)
* High risk of hemorrhage - where fluid volume expansion is planned prior to delivery (e.g. placenta previa, placenta accreta)

Exclusion Criteria:

* Starting BP is less than 100 systolic: as the lower limit for intervention defined in this study is 90sys which will likely be within the error of the BP measurement device
* There is a prolonged (more than 2 hour) wait between testing and spinal insertion: as patients may become more dehydrated affecting hypotension rates

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy women who are admitted to the hospital for a scheduled elective cesarean delivery
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Passive leg raise related cardiac output change and correlation with presence of phenylephrine infusion resistant hypotension | One hour prior to scheduled cesarean delivery
Passive leg raise related plethysmography variability index change and correlation with presence of phenylephrine infusion resistant hypotension | One hour prior to scheduled cesarean delivery

SECONDARY OUTCOMES:
Baseline plethysmography variability index, plethysmography index and systemic vascular resistance values and correlation with presence of phenylephrine infusion resistant hypotension | From administration of spinal anesthetic to delivery of infant
Passive leg raise related plethysmography variability index and cardiac output change and correlation with severe phenylephrine resistant hypotension | One hour prior to scheduled cesarean delivery
  Defined as requirement of 3 or more rescue bolus doses of vasopressor/anticholinergic according to intervention protocol
Passive leg raise related plethysmography variability index and cardiac output change and correlation with hypotension associated with bradycardia | One hour prior to scheduled cesarean delivery
Presence of phenylephrine infusion associated side effects | From administration of spinal anesthetic to delivery of infant
  Hypertension or normotensive bradycardia associated with phenylephrine infusion use
Presence of recurrent (3 or more) episodes of phenylephrine infusion associated side effects | From administration of spinal anesthetic to delivery of infant
Maternal cardiac output and systemic vascular resistance changes following spinal anesthesia | From administration of spinal anesthesia to delivery of infant
Umbilical cord gases | At delivery of infant
Apgar scores at 1 and 5 minutes | At delivery of infant

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Women's Hospital, Vancouver, British Columbia, Canada